CLINICAL TRIAL: NCT07365514
Title: Blackcurrants Mitigate Postmenopausal Bone Loss Through Gut Microbiota-Bone Axis: A Randomized Clinical Trial Coupled With a Multi-Omics Approach to Inform Precision Nutrition
Brief Title: Blackcurrants Modify Gut Microbiota and Reduce Osteoporosis Risk in Postmenopausal Females
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Ock Chun, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B2025-0380; 2025-67018-45103 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal Osteoporosis; Gut Microbiome; Menopause
Keywords: blackcurrant; gut microbiome; osteoporosis; menopause; females; bone aging
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of three groups and asked to consume three capsules per day in the morning for 12 months as follows: 1) 3 capsules containing 784 mg blackcurrant (BC) extract (261.33 mg BC and 130.67 mg placebo per capsule; low BC group); or 2) 3 capsules containing 1,176 mg BC extract (three 392 mg BC capsules; high BC group); or 3) 3 placebo capsules (392 mg placebo per capsule; control group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-BC Group (Active Comparator): Low-dose BC extract
  Interventions: Drug: Blackcurrant (BC) extract
- High-BC Group (Active Comparator): High-dose BC extract
  Interventions: Drug: Blackcurrant (BC) extract
- Control Group (Placebo Comparator): Placebo (no BC extract)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blackcurrant (BC) extract — Consume three capsules per day containing 784 mg of blackcurrant (BC) extract (261.33 mg BC and 130.67 mg placebo per capsule)
  Arms: Low-BC Group
Drug: Blackcurrant (BC) extract — Consume three capsules containing 1,176 mg BC of extract (392 mg BC per capsule)
  Arms: High-BC Group
Drug: Placebo — Consume three placebo capsules (392 mg placebo per capsule)
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of blackcurrant (BC) supplementation on changes in bone density and gut microbiome composition in postmenopausal females.

DETAILED DESCRIPTION:
Postmenopausal osteoporosis (PMO) is a debilitating and progressive metabolic bone disorder caused by estrogen deficiency after menopause, leading to an imbalance in bone remodeling. Owing to its high morbidity and serious complications, substantial efforts have been devoted to its prevention and treatment. Emerging evidence indicates that the gut microbiome plays a pivotal role in bone health through immune and endocrine pathways, influencing bone turnover via cytokine signaling, metabolite production, and calcium balance.

Our previous 6-month trial suggested that blackcurrant (BC) may exert bone-protective effects through integrated effects on bone remodeling, gut microbiota, and metabolite signaling. Therefore, the overall goal of this study is to investigate the effects of BC supplementation on changes in gut microbiota and bone density in postmenopausal females and to elucidate the interrelationship of BC and gut microbiota with regard to bone loss mitigation. This will be accomplished using a multidisciplinary, comprehensive multi-omics approach to examine interactions among BC, gut microbiota, bacterial metabolites, and the immune and endocrine systems in relation to bone metabolism.

Investigators will conduct a randomized, placebo-controlled trial of BC supplementation for 12 months in postmenopausal females aged 45-70 years. The primary endpoint will be changes in whole-body, lumbar spine, total hip, and femoral neck bone mineral density. The secondary endpoint will be changes in biomarkers of bone remodeling. To further delineate underlying mechanisms, changes in the community structure of the gut microbiome, inflammatory-immune markers, and endocrine markers will be assessed. Additional analyses will include proteomics to identify protein biomarkers, metabolomics to identify key metabolites associated with BC supplementation and bone-related outcomes, and genotyping to evaluate genetic polymorphisms in bone-related genes.

The specific objectives of this study are to investigate the effects of BC extract on: 1) bone density and bone remodeling biomarkers; and 2) changes in gut microbiota abundance and composition, inflammatory-immune and endocrine biomarkers, protein biomarkers (proteomics), key metabolites (metabolomics), and their relationships with changes in bone density, including evaluation of genetic polymorphisms in bone-related genes (genomics).

This study will provide further insight into whether and how BC consumption may reduce the risk of postmenopausal bone and will improve understanding of the role of the gut microbiome in postmenopausal bone loss. Findings may provide novel insight into how anthocyanin-rich berries reduce PMO risk via the gut-bone axis and may support the development of future dietary recommendations and strategies for adult females approaching or experiencing menopause.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal (defined as no more than 10 years since final menstrual cycle) females aged 45-70 years
* not on hormone replacement therapy for at least one year before initiation of the study
* maintaining normal exercise level (< 7 hours/week) and willing to avoid exercise for 24 hours prior to blood and stool sampling
* willing to ingest a dietary blackcurrant supplement or placebo (up to 1,176 mg/day, three 392mg capsules)
* willing to avoid other dietary supplements for the duration of the study
* willing to avoid intake of foods extremely rich in anthocyanins and fermented dairy products containing viable Bifidobacteria or Lactobacilli
* willing to have three blood draws, three stool collections, and three bone scans

Exclusion Criteria:

* history of cardiovascular disease, osteoporosis, metabolic bone disease, cancer, diabetes mellitus, arthritis, or other chronic inflammatory diseases
* current smokers
* taking prescription medications known to alter bone and calcium metabolism
* taking anabolic agents such as parathyroid hormone or growth hormone, or steroid within 3 months before the start of the study
* taking medications that alter bleeding (such as antiplatelets or anticoagulants) or those with a bleeding disorder
* alcohol consumption exceeding 2 drinks/day (approximately 14g of ethanol per drink) or a total of 12/week
* those with planned surgery during the study period or within 2 weeks of ending the intervention
* those with sensitivities or allergies to any of the ingredients for the placebo (rice powder)
* planning a procedure that includes iodine, barium or nuclear medicine isotopes within the study period
* UConn students and/or employees who any key personnel teach or who report to any key personnel
* study key personnel, partners of key personnel, or dependents/relatives of any key personnel

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal females
Enrollment: 159 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | From baseline to months 6 and 12
  Changes from baseline in whole-body, lumbar spine, total hip and femoral neck BMD at months 6 and 12 measured via dual energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Serum markers of bone remodeling | From baseline to months 6 and 12
  Changes in serum concentrations of bone remodeling markers including procollagen type I N-propeptide (P1NP), bone alkaline phosphatase (BALP), receptor activator of nuclear factor kappa-Β ligand (RANKL), and collagen Type I C-Telopeptide (CTX1)

OTHER OUTCOMES:
Changes in community structure of gut microbiota | from baseline to months 6 and 12
  Changes in gut microbial composition will be assessed using alpha diversity (species richness and Shannon diversity) and beta diversity metrics, including Bray-Curtis dissimilarity (community abundance) and Jaccard distance (presence/absence). Taxonomic composition will be compared between groups by evaluating relative abundance at the genus and phylum levels.
Plasma inflammatory-immune markers | from baseline to months 6 and 12
  Inflammatory biomarkers will be assessed in plasma, including IL-1beta and TNF-alpha. Additional immune response markers related to T helper cell subtypes (Th1, Th2, Th17) will be measured in plasma (e.g., interleukin (IL)-2, IL-4, IL-6, IL-10, TNF, IL-17A). CD4+ Th17 and regulatory T cell (Treg) responses will also be evaluated from peripheral blood mononuclear cells (PBMCs).
Plasma endocrine markers | from baseline to months 6 and 12
  Changes in plasma concentrations of endocrine markers including insulin-like growth factor-1 (IGF-1) and cyclic glycine-proline (cGP)
Omics outcomes | from baseline to months 6 and 12
  Metabolomics, proteomics, and genotyping will be performed to identify biomarkers associated with blackcurrant supplementation and bone-related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ock Chun, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Department of Nutritional Sciences, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Once research proceedings and manuscripts are published, we will make our results available to both the community of scientists interested in postmenopausal osteoporosis and those studying the biology of inflammation-induced bone resorption and avoid unintentional duplication of research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Unlimited time after papers are published.
Access Criteria: Our plan for sharing of data generated by this project includes the following:
  1. Presentations at national scientific meeting. From the project, it is expected that approximately two presentations at national meetings would be appropriate.
  2. Publication in peer-reviewed journals. It is our explicit intention that the study findings and key data will be placed in a readily accessible public database. All efforts will be made to rapidly release data through publication of results as quickly as possible following our analysis of experiment data. Data used in publications will be released in a timely manner.